CLINICAL TRIAL: NCT03649919
Title: Multi-center Clinical Study on the Diagnosis and Treatment Management of Rare Neurological Disease in Children
Status: Withdrawn | Type: Observational
Why Stopped: lack of funding
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Children's Medical Center (Other); Xinhua Hospital of Shanghai Jiaotong University (Unknown)
Responsible Party: Sponsor
Other Study IDs: EKYY-MCSDTMRNDC
Record Dates: First submitted 2018-08-26; First posted 2018-08-28 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Xlsma; DMD; X-ALD; TSC
MeSH Terms: conditions — Arthrogryposis multiplex congenita, distal, X-linked; Adrenoleukodystrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1 spinal muscular atrophy, SMA: Progressive muscular atrophy (SMA) is a group of autosomal recessive neuromuscular diseases characterized by degeneration of the anterior horn cells of the spinal cord, which is characterized by progressive generalized muscle weakness and muscle atrophy. The incidence of SMA is about 1/11000, and the occurrence of SMA is caused by mutation of the SMN1 gene. SMA can be classified into type I-III according to age of onset, maximum muscle activity, and survival.
- 2 DMD: Progressive muscular dystrophy (DMD) is a group of hereditary skeletal muscle degeneration diseases. It is clinically characterized by slow and progressive development of muscle atrophy and muscle weakness. The inheritance can be divided into sexual chain recessiveness. Genetic type. For children with high suspected DMD/BMD, the current DMD diagnosis is preferred by MLPA method for detection of DNA in peripheral blood; MLPA diagnostic kit can only detect about 65% of large gene deletions or repeat types, thus detecting undetected gene mutations.
- 3 X-linked adrenoleukodystrophy X-ALD: X-linked adrenoleukodystrophy X-ALD is an X-linked episode of a group of diseases characterized by progressive central nervous system demyelination and adrenal insufficiency. About 1/20000 male children. Most cases of X-ALD are treated for neurological symptoms for the first time, most of them start from 3-10 years old. Early manifestations include slow mental function, decreased academic performance, lack of interest or hyperactivity, difficulty in speech, difficulty in articulation, etc. Visual impairment and progressive hemiplegia are more common symptoms.
- 4 tuberous sclerosis complex，TSC: Tuberous sclerosis complex (TSC) is an autosomal dominant genetic disease involving multiple systems. About 1 in every 6,000-10,000 people in TSC suffer from tuberous sclerosis, and children in the neurology department are diagnosed with developmental delay or seizures, and about 2/3 have no positive family history. Nearly 2 million people worldwide suffer from TSC, and there are about 200,000 in China.

INTERVENTIONS:
Other:  — Patients receive routine diagnostic and treatment medications.

SUMMARY:
The incidence of rare diseases is extremely low, the disease is numerous, the symptoms are serious, and the detection technology is complicated. Countries have different definitions of rare diseases. The definition of rare diseases in China is defined as: diseases with a prevalence of less than 1 in 500 000 or newborns with an incidence of less than 1/10 000 are rare diseases. Due to the low incidence of rare diseases and the accumulation of multiple organs and systems in most diseases, clinicians lack comprehensive and systematic understanding. Patients often face great difficulties in seeking medical treatment and diagnosis. Currently, there is a lack of systematic and rare diseases in China. Management, diagnosis and treatment of rare diseases, making the diagnosis of rare diseases, prevention interventions seriously lagging behind, obviously behind the management of developed countries and regions; rare diseases are mostly related to genetic variation, with the clinical application of genetic diagnosis technology, more and more Many genetically related rare diseases have been diagnosed at an early stage; at present, precision medicine is rapidly developing, and more and more rare disease clinical trials have entered the country, bringing prospects for the treatment of rare diseases. For this reason, the management of rare diseases is particularly important.

At present, some rare diseases of the nervous system can be treated early; for example, immune-related rare diseases have common normative immunotherapy and functional disability prevention, and the characteristics of single disease management of each disease; hereditary degenerative rare diseases such as progressive 2-3 multi-center clinical trials of spinal muscular atrophy and progressive muscular dystrophy have been entered into our hospital (in our hospital), X-linked pre-diagnosis of adrenal malnutrition genetic diseases, and appropriate treatment time is selected. Stem cell transplantation is in research and planning; the long-term management and comprehensive treatment of nodular sclerosis and Dravet syndrome are important for the prevention and treatment of diseases; therefore, the early diagnosis, pathogenesis and standardized treatment of rare diseases of the nervous system are urgent. And necessity.

ELIGIBILITY:
1. SMA:

Inclusion criteria: patients meet the all the following criteria:

1. Clinically manifestation: hypotonia, progressive symmetric and proximal weakness affecting the legs more than the arms, sparing of the facial muscles but often with bulbar muscle weakness.
2. Neurogenic EMG. EMG is also usually not needed in type 1 and 2 children; this investigation can help in more chronic forms in which the phenotype might be less striking.
3. Along with EMG and NCV test, a muscle or nerve biopsy can be used to diagnose spinal muscular atrophy if molecular genetic testing of SMN1 does not identify mutations.
4. Genetic testing of SMN1/SMN2: Homozygous absence of exons 7 and 8 of the SMN1 gene(96%), or only of exon 7, or other mutations. SMN2 copy numbers may vary. Genetic testing is the gold standard of diagnosis.

Exclusion Criteria: None.

-

2. DMD:

Inclusion criteria: patients meet the all the following criteria:

1. Clinically manifestation: weakness, clumsiness, a Gowers' sign, difficulty with stair climbing, or toe walking. developmental delay or increased concentrations of serum enzymes such as alanine aminotransferase, aspartate aminotransferase, lactate dehydrogenase, or very high creatine kinase level.
2. Dystrophin gene mutation: dystrophin gene deletion and duplication testing is usually the first confirmatory test best done by MLPA or comparative genomic hybridisation array. Approximately 70% of individuals with DMD have a single-exon or multi-exon deletion or duplication in the dystrophin gene. If deletion or duplication testing is negative, genetic sequencing should be done to screen for the remaining types of mutations that are attributed to DMD (approximately 25-30%).
3. Muscle biopsy: if genetic testing does not confirm a clinical diagnosis of DMD, then a muscle biopsy sample should be tested for the presence of dystrophin protein by immunohistochemistry of tissue cryosections or by western blot of a muscle protein extract. Muscle samples from DMD patient has no dystrophin present, while BMD Becker muscular dystrophy (with some partially functional dystrophin present).

Exclusion Criteria: None. -

3. X-ALD:

Inclusion criteria: patients meet the all the following criteria:

1. Clinically manifestation:

1. Attention deficit disorder or hyperactivity; progressive impairment of cognition, behavior, vision, hearing, and motor function follow the initial symptoms and often lead to total disability within six months to two years.
2. Adrenomyeloneuropathy (AMN) manifests as progressive stiffness and weakness of the legs, sphincter disturbances, sexual dysfunction, and often, impaired adrenocortical function; all symptoms are progressive over decades, most commonly in an individual in his twenties or middle age.
3. Magnetic resonance imaging shows cerebral demyelination.

2. Dystrophin gene mutation: The diagnosis of X-ALD is usually established in a female proband with detection of a heterozygous ABCD1 pathogenic variant and elevated VLCFA.

Exclusion Criteria: None. -

4. TSC:

Inclusion criteria:patients meet the all the following criteria:

A. Clinical diagnostic criteria:

1. Major features: (1) Hypomelanotic macules (≥3, at least 5-mm diameter). (2) Angiofibromas (≥3) or fibrous cephalic plaque. (3) Ungual fibromas (≥2). (4) Shagreen patch. (5) Multiple retinal hamartomas. (6) Cortical dysplasias. (7) Subependymal nodules. (8) Subependymal giant cell astrocytoma. (9) Cardiac rhabdomyoma. (10) Lymphangioleiomyomatosis (LAM). (11) Angiomyolipomas (≥2).
2. Minor features: (1)"Confetti" skin lesions. (2) Dental enamel pits (>3). (3) Intraoral fibromas (≥2). (4) Retinal achromic patch. (5) Multiple renal cysts. (6) Nonrenal hamartomas.

Two major features or one major feature with ≥2 minor features can diagnose. Either one major feature or ≥2 minor features can diagnosis possibly.

B. Genetic diagnostic criteria:

The identification of either a TSC1 or TSC2 pathogenic mutation in DNA from normal tissue is sufficient to make a definite diagnosis of TSC.

Exclusion Criteria: None.

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient affected with Xlsma, DMD, X-ALD or TSC aged frome 0 to 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
spinal muscular atrophy, SMA | from birth, to 18 years old
  Diagnosed based on the clinical criteria and genetic analysis. The details clinical diagnosis refer to the inclusion criteria. The genetic diagnosis of a Spinal Muscular Atrophy is established in a patient by identification of a homozygous absence of SMN1 exon 7 using SMA MLPA test (MRC-holland P021-A2).
DMD | from birth, to 18 years old
  Diagnosed based on the clinical criteria and genetic analysis. The details clinical diagnosis refer to the inclusion criteria. The genetic diagnosis of a Dystrophinopathy is established in a male patient by identification of a hemizygous pathogenic variant (including exon or whole-gene deletions/duplications, intragenic deletions/insertions, missense, nonsense, and splice site variants) in DMD gene using a multigene panel sequencing test (Agilent ClearSeq Inherited Disease panel kit).
X-linked adrenoleukodystrophy X-ALD | from birth, to 18 years old
  Diagnosed based on the clinical criteria and the details clinical diagnosis refer to the inclusion criteria.
tuberous sclerosis complex，TSC | from birth, to 18 years old
  Diagnosed based on the clinical criteria and genetic analysis. The details clinical diagnosis refer to the inclusion criteria. The genetic diagnosis of a TSC is established in a patient by identification of a heterozygous pathogenic variant (including exon or whole-gene deletions, intragenic deletions/insertions, missense, nonsense, and splice site variants) in TSC1 or TSC2 using a multigene panel sequencing test (Agilent ClearSeq Inherited Disease panel kit).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes